CLINICAL TRIAL: NCT01239394
Title: Phase II Trial Ofatumumab for Initial Systemic Treatment of Indolent B-cell Lymphoma
Brief Title: Ofatumumab for Initial Systemic Treatment of Indolent B-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Beth Israel Deaconess Medical Center (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Jeremy Abramson, MD, Director, Lymphoma Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-271
Record Dates: First submitted 2010-11-10; First posted 2010-11-11 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-09

CONDITIONS: Follicular Lymphoma; Marginal Zone Lymphoma; Small Lymphocytic Lymphoma
Keywords: NHL; ofatumumab
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ofatumumab (Other): single-arm, open-label, interventional
  Interventions: Drug: ofatumumab

INTERVENTIONS:
Drug: ofatumumab — Weekly infusion for 8 weeks
  Other Names: GSK1841157; HuMax-CD20

SUMMARY:
Ofatumumab is a drug that works by attaching to the CD20 molecule found on the surface of cancerous B cells, and then triggering the death of those cells. It is approved by the FDA for treatment of another B-cell cancer, chronic lymphocytic leukemia, and also has evidence of success in people who's B-cell lymphomas have relapsed after initial treatments. In this research study we are looking to see if ofatumumab is effective and safe in treating previously untreated B-cell NHL.

DETAILED DESCRIPTION:
* Participants will receive ofatumumab once a week for 8 weeks by intravenous infusion (Days 1, 8, 15, 22, 29, 36, 43, and 50).
* Participants will be seen weekly during the 8 week treatment period and will have the following tests and procedures performed: Blood tests, performance status and physical examination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed indolent CD20+B-cell NHL of the following histologies: follicular lymphoma, grades 1-2; Marginal zone lymphoma (extranodal, nodal or splenic); small lymphocytic lymphoma; low-grade B-cell lymphoma not otherwise specified with CD20+ expression
* Measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension as 20mm or greater CT scan or MRI
* No previous chemotherapy, antibody therapy or radioimmunotherapy for this disease. Patients previously treated with external beam radiation alone are eligible
* 18 years of age or older
* Life expectancy of greater than 3 months
* ECOG Performance status of 0, 1 or 2
* Organ function as described in the protocol
* Women of child-bearing potential and men must agree so use adequate contraception prior to study entry and for the duration of study participation

Exclusion Criteria:

* Prior chemotherapy, antibody therapy or radioimmunotherapy for lymphoma
* Participants may not be receiving any other investigational agent
* Participants with known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ofatumumab
* Prior exposure to ofatumumab or other targeted anti-CD20 therapies including rituximab
* Known HIV positivity
* Positive serology for Hepatitis B
* Positive serology for Hepatitis C
* Participants who are candidates for curative radiotherapy, unless radiation therapy is considered too toxic (as in abdominal disease), or is refused by the patient
* New York Heart Association Classification III of IV heart disease
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection that is not optimally treated with antibiotics, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women
* History of a different malignancy are ineligible except for the following circumstances: Individuals with a history of other malignancy are eligible if they have been disease-free for at least one year and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible even if diagnosed and treated within the past 1 year: localized prostate cancer, prostate cancer with elevated PSA but no measurable disease on CT scans or bone scan, cervical cancer in situ, breast ductal carcinoma in situ and non-melanoma skin cancers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy S. Abramson, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The number enrolled (43) and number starting study (42) do not match because one patient never began study treatment due to an acute stroke prior to any study treatment.
Period: Overall Study
Arm/Group | Ofatumumab
Started | 42
Completed | 41
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 64.4 [33.7 to 91.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 36
  More than one race | 2
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 42
Lymphoma type [Count of Participants; unit: Participants]
  Follicular | 28
  Marginal zone | 4
  Small lymphocytic | 10

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Complete Response Rate (CRR)
Description: Evaluate clinical efficacy of ofatumumab in previously untreated indolent B-cell lymphomas, as measured by complete response rate (CRR).
  Complete response = all previously enlarged fluorodeoxyglucose (FDG)-avid or positron emission tomography (PET)-positive lymph nodes regressed to normal size (<=1.5 cm in greatest diameter)
Time Frame: 1-month post-treatment
Measure: Number; unit: percentage of patients
Arm/Group | Ofatumumab
Number analyzed (Participants) | 41
percentage of patients | 9.5

2. Secondary Outcome: Overall Response Rate (ORR)
Description: Evaluate clinical efficacy of ofatumumab in previously untreated indolent B-cell lymphomas, as measured by overall response rate (ORR).
  Overall response = Complete response (CR) + Partial response (PR) CR = all previously enlarged fluorodeoxyglucose (FDG)-avid or positron emission tomography (PET)-positive lymph nodes regressed to normal size (<=1.5cm in greatest diameter) PR = >=50% decrease in SPD of up to six largest dominant masses, no increase in size of other nodes; FDG avid or PET positive before therapy, one or more nodes PET positive at previously involved site, or variably FDG avid or PET negative with regression at CT
Time Frame: 1-month post-treatment
Measure: Number; unit: percentage of patients
Arm/Group | Ofatumumab
Number analyzed (Participants) | 41
percentage of patients | 52

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Percentage of patients with progression-free survival during 12 months post-treatment progression-free survival: patients live with the disease, but it does not get worse
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Ofatumumab
Number analyzed (Participants) | 41
percentage of patients | 86 [72 to 99]

4. Secondary Outcome: Toxicity: Infusion Reactions, Grade 3-4 Infections, and Neutropenia
Description: Evaluate safety of ofatumumab monotherapy in this patient population Toxicities are graded 1 (mild), 2 (moderate), 3 (severe), and 4 (life-threatening)
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Ofatumumab
Number analyzed (Participants) | 42
Participants
  Infusion reactions (grade 1-2) | 22
  Infusion reactions (grade 3) | 7
  Infections (grade 3-4) | 1
  Neutropenia (grade 3-4) | 0

ADVERSE EVENTS:
Arm/Group | Ofatumumab
Serious Adverse Events (participants affected / at risk) | 2/42
Other Adverse Events (participants affected / at risk) | 38/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ofatumumab (N=42)
Vestibular Schwannoma (Nervous system disorders) | 1 (1) — Grade 2, unrelated
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 4, expected and unrelated
Fever (General disorders) | 1 (1) — Grade 2, expected and unrelated
Headache (Nervous system disorders) | 1 (1) — grade 3, expected and unrelated
Photophobia (Eye disorders) | 1 (1) — Grade 2, unexpected and unrelated
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ofatumumab (N=42)
Allergic reaction (Immune system disorders) | 28 (30)
Fatigue (General disorders) | 19 (21)
Nausea (Gastrointestinal disorders) | 9 (12)
Headache (Nervous system disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 6 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Infusion related react (General disorders) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 5 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 5 (5)
Platelet count decrease (Investigations) | 5 (5)
Anemia (Blood and lymphatic system disorders) | 4 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Blood bilirubin increase (Investigations) | 4 (4)
Constipation (Gastrointestinal disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Skin and subcutaneous (Skin and subcutaneous tissue disorders) | 4 (4)
Alanine aminotransferase (Investigations) | 3 (5)
Anxiety (Psychiatric disorders) | 3 (3)
Bladder infection (Infections and infestations) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Neutrophil count decrease (Investigations) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No